CLINICAL TRIAL: NCT00147576
Title: Randomized, Placebo-Controlled Parallel Group Study Comparing Effect Of Three Doses Of CP-866,087 And Naltrexone On Acute Alcohol Consumption And Craving After Seven Days Of Treatment In Alcohol Dependent (DSM IV) Subjects Who Are Not Currently Seeking Treatment
Brief Title: Study To Examine Effect Of CP-866,087 On Consumption And Craving Of Alcohol In Alcohol Dependent Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5051005
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — CP-866,087

INTERVENTIONS:
Drug: CP-866,087

SUMMARY:
Test the hypothesis that increasing doses of CP-866,087 will decrease the total number of drinks consumed during a 2 hour acute alcohol consumption assessment and to determine the safety and tolerability of multiple doses of CP-866,087 in alcohol dependent subjects compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the DSM-IV criterion for current alcohol dependence.
* Subject is currently not engaged in, and does not want, treatment for alcohol related problems.

Exclusion Criteria:

* Subject meets criteria for current DSM-IV diagnosis for any other psychoactive substance abuse or dependence disorder, excluding nicotine and caffeine.
* Specialized inpatient or outpatient alcoholism or other addiction treatment (except nicotine) within the past 12 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-12; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The amount of alcohol consumed will be based on the total number of standardized drinks consumed during a two-hour laboratory-based self-administration procedure following 7 days of treatment with study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Lenexa, Kansas
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, San Antonio, Texas